CLINICAL TRIAL: NCT03856723
Title: Predicting Outcomes of Cardiac Surgery-associated Acute Kidney Injury Using Biomarkers At Initiation of REnal Replacement Therapy (POCKET)
Brief Title: Predicting Outcomes of Cardiac Surgery-associated Acute Kidney Injury Using Biomarkers At Initiation of RRT
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: POCKET
Record Dates: First submitted 2019-02-23; First posted 2019-02-27 (Actual); Last update posted 2022-06-01 (Actual); Status verified 2022-05

CONDITIONS: Acute Kidney Injury
Keywords: Acute Kidney Injury; Renal Replacement Treatment; Biomarker
MeSH Terms: conditions — Acute Kidney Injury | interventions — Renal Replacement Therapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 90 Days
Biospecimen Retention: Samples With DNA — Blood samples are drawn before the first dialysis session after post cardiac surgery associated AKI ( initializing RRT). Blood is drawn into Vacutainer tubes containing EDTA, and immediately placed on ice and centrifuged within 1 h. All the samples are stored at -70°C until analysis.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Renal Replacement Therapy — Indications for RRT were defined as previously reported.
  1. Kidney Disease: Improving Global Outcomes (KDIGO) stage 2 ;
  2. severe sepsis, persistence of hypotension (for more than 6 h) despite preload optimization and use of vasopressors or catecholamines (norepinephrine or epinephrine >0.1 μg/kg/min),
  3. refractory fluid overload (worsening pulmonary edema, PaO2/FiO2 <300 mm Hg or fluid balance >10% of body weight),
  4. low probability of rapid renal recovery according to the judgment of the intensivists and nephrologists.

SUMMARY:
The aim of this study was to verify the prognostic value of functional kidney biomarkers on survival and renal function recovery in cardiac surgery patients with acute kidney injury.

DETAILED DESCRIPTION:
Cardiac surgery-associated acute kidney injury (CSA-AKI) is the second most common type of AKI after septic AKI and is associated with increased mortality and morbidity. Few biomarkers were validated as outcome-specific biomarkers in patients developing AKI after cardiac surgery at initiation of RRT. This study was designed to not only verify the prognostic value of functional kidney biomarkers on survival, but also predict it severity in order to optimize clinical decision making with respect to dialysis initiation and discontinuation.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing cardiac surgery who required renal replacement therapy.

Exclusion Criteria:

* History of End Stage Renal Disease or on Dialysis
* prior kidney transplantation
* patients with a DNR order or "do not escalate care" order

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The incidence of cardiac surgery-associated AKI (CSA-AKI) varies from 5% to 42%. CSA-AKI is the second most common cause of AKI in the intensive care setting (after sepsis) and is independently associated with increased morbidity and mortality.
Sampling Method: Probability Sample
Enrollment: 1200 (Estimated)
Dates: Start 2019-03-01 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
28-day mortality | 28 days
  Death from any cause at 28 days
Dependence on renal-replacement therapy at 28 days in survivors | 28 days
  Dependence on renal-replacement therapy was defined as surviving dependent on RRT

SECONDARY OUTCOMES:
60- and 90-day mortality | Up to 60 or 90 days
  Death from any cause at 60- and 90-days
Length of stay in the ICU | Up to 90 days or ICU discharge
  the length of stay in the ICU
Length of stay in the hospital | Up to 90 days or hospital discharge
  the length of stay in the hospital
Adverse events | Up to 90 days
  with a focus on the complications potentially related to acute kidney injury or renal-replacement therapy during the first 7 days after enrollment
the number of days free of renal-replacement therapy, mechanical ventilation at 28 days | 28 days
  the number of days free of renal-replacement therapy, mechanical ventilation at 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Zhe Luo, PhD, Study Chair — Fudan University
Locations (1):
- Zhongshan hospital, Fudan university, Shanghai, China